CLINICAL TRIAL: NCT02526043
Title: A Prospective Randomized Control Trail of Laparoscopic Versus Open Liver Resection for Hepatocellular Carcinoma
Brief Title: Laparoscopic Versus Open Liver Resection for Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Lunxiu Qin, Department of general surgery, Huashan hospital, Fudan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Huashan 002
Record Dates: First submitted 2015-08-05; First posted 2015-08-18 (Estimated); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- laparoscopic hepatectomy (Experimental): The HCC patients who meet the Louisville consensus will be underwent the liver resection by laparoscopic surgery
  Interventions: Procedure: laparoscopic hepatectomy
- Open hepatectomy (Experimental): The HCC patients who meet the Louisville consensus will be underwent the liver resection by open surgery
  Interventions: Procedure: Open hepatectomy

INTERVENTIONS:
Procedure: laparoscopic hepatectomy — The HCC patients who meet the Louisville consensus will underwent liver resection by laparoscopy
  Arms: laparoscopic hepatectomy
Procedure: Open hepatectomy — The HCC patients who meet the Louisville consensus will underwent liver resection by open surgery
  Arms: Open hepatectomy

SUMMARY:
The purpose of the study is to observe the curative effect and safety of laparoscopic versus open liver resection for hepatocellular carcinoma.

DETAILED DESCRIPTION:
Liver resection is the most important treatment of hepatocellular carcinoma (HCC). Open hepatectomy was regarded as a giant surgery because of its big incision, influence of the liver function, and long hospital stay. Laparoscopic hepatectomy was widely used since it was reported by Reich in 1991. With the constant innovation of laparoscopic technique and equipment, there is no penalty area in laparoscopic hepatectomy. The Louisville consensus proposed that the best indication for laparoscopic hepatectomy was the tumor diameter < 5cm, located in segment II-VI.

Previous studies shows that compared with the open surgery, laparoscopic hepatectomy has the advantages of shorter operation time, less bleeding, shorter hospitalization time. The mortality, mobility, the overall survival and the disease-free survival was same in these two groups.

So far, however, the curative effect and safety research of laparoscopic versus open liver resection for HCC is limited to retrospective study and case-control study. A prospective, randomized, controlled study is urgently needed.

This study was proceeded to observe the curative effect and safety of laparoscopic versus open liver resection for HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis was HCC
2. The tumor was located in segment: II, III, IVb, V, VI
3. The tumor diameter < 5cm
4. Without thrombosis in the portal vein, hepatic vein or bile duct
5. Without intrahepatic and systemic metastasis
6. The Child-pugh score was A-B7
7. The ASA（American Society of Anesthesiologists） score was I-III
8. The patient age was between 18-75
9. Sign the informed consent, and can fully understand the research content

Exclusion Criteria:

1. Have surgery contraindications
2. Pregnant or lactating women
3. The Child-pugh score was B8-C
4. The ASA（American Society of Anesthesiologists） score was IV-V
5. With other malignant tumor
6. With mental illness
7. Participated in other clinical trials in the last three months
8. Underwent other treatments(chemotherapy or radiotherapy) before operation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-08; Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The overall survival of HCC patients after operation

SECONDARY OUTCOMES:
Disease free survival | 5 years
  The disease free survival of HCC patients after operation
Incidence of postoperative complications | 1 month
  Incidence of postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Lunxiu Qin, MD, Principal Investigator — Department of general surgery, Huashan hospital, Fudan University
Locations (1):
- Huashan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ishizawa T, Gumbs AA, Kokudo N, Gayet B. Laparoscopic segmentectomy of the liver: from segment I to VIII. Ann Surg. 2012 Dec;256(6):959-64. doi: 10.1097/SLA.0b013e31825ffed3. PMID 22968066
- [Background] Reich H, McGlynn F, DeCaprio J, Budin R. Laparoscopic excision of benign liver lesions. Obstet Gynecol. 1991 Nov;78(5 Pt 2):956-8. PMID 1833688
- [Background] Chen KH, Jeng KS, Huang SH, Chu SH. Laparoscopic caudate hepatectomy for cancer--an innovative approach to the no-man's land. J Gastrointest Surg. 2013 Mar;17(3):522-6. doi: 10.1007/s11605-012-2115-z. Epub 2013 Jan 8. PMID 23297026
- [Background] Buell JF, Cherqui D, Geller DA, O'Rourke N, Iannitti D, Dagher I, Koffron AJ, Thomas M, Gayet B, Han HS, Wakabayashi G, Belli G, Kaneko H, Ker CG, Scatton O, Laurent A, Abdalla EK, Chaudhury P, Dutson E, Gamblin C, D'Angelica M, Nagorney D, Testa G, Labow D, Manas D, Poon RT, Nelson H, Martin R, Clary B, Pinson WC, Martinie J, Vauthey JN, Goldstein R, Roayaie S, Barlet D, Espat J, Abecassis M, Rees M, Fong Y, McMasters KM, Broelsch C, Busuttil R, Belghiti J, Strasberg S, Chari RS; World Consensus Conference on Laparoscopic Surgery. The international position on laparoscopic liver surgery: The Louisville Statement, 2008. Ann Surg. 2009 Nov;250(5):825-30. doi: 10.1097/sla.0b013e3181b3b2d8. PMID 19916210
- [Background] Afaneh C, Kluger MD. Laparoscopic liver resection: lessons at the end of the second decade. Semin Liver Dis. 2013 Aug;33(3):226-35. doi: 10.1055/s-0033-1351780. Epub 2013 Aug 13. Danish, English. PMID 23943103
- [Result] Bryant R, Laurent A, Tayar C, Cherqui D. Laparoscopic liver resection-understanding its role in current practice: the Henri Mondor Hospital experience. Ann Surg. 2009 Jul;250(1):103-11. doi: 10.1097/SLA.0b013e3181ad6660. PMID 19561476
- [Result] Topal B, Fieuws S, Aerts R, Vandeweyer H, Penninckx F. Laparoscopic versus open liver resection of hepatic neoplasms: comparative analysis of short-term results. Surg Endosc. 2008 Oct;22(10):2208-13. doi: 10.1007/s00464-008-0023-9. Epub 2008 Jul 12. PMID 18622562
- [Result] Tranchart H, Di Giuro G, Lainas P, Roudie J, Agostini H, Franco D, Dagher I. Laparoscopic resection for hepatocellular carcinoma: a matched-pair comparative study. Surg Endosc. 2010 May;24(5):1170-6. doi: 10.1007/s00464-009-0745-3. Epub 2009 Nov 14. PMID 19915908
- [Result] Cai XJ, Yang J, Yu H, Liang X, Wang YF, Zhu ZY, Peng SY. Clinical study of laparoscopic versus open hepatectomy for malignant liver tumors. Surg Endosc. 2008 Nov;22(11):2350-6. doi: 10.1007/s00464-008-9789-z. Epub 2008 Feb 23. PMID 18297354
- [Result] Dagher I, Lainas P, Carloni A, Caillard C, Champault A, Smadja C, Franco D. Laparoscopic liver resection for hepatocellular carcinoma. Surg Endosc. 2008 Feb;22(2):372-8. doi: 10.1007/s00464-007-9487-2. Epub 2007 Aug 18. PMID 17704878
- [Result] Lee KF, Chong CN, Wong J, Cheung YS, Wong J, Lai P. Long-term results of laparoscopic hepatectomy versus open hepatectomy for hepatocellular carcinoma: a case-matched analysis. World J Surg. 2011 Oct;35(10):2268-74. doi: 10.1007/s00268-011-1212-6. PMID 21842300
- [Result] Slim A, Garancini M, Di Sandro S, Mangoni I, Lauterio A, Giacomoni A, De Carlis L. Laparoscopic versus open liver surgery: a single center analysis of post-operative in-hospital and post-discharge results. Langenbecks Arch Surg. 2012 Dec;397(8):1305-11. doi: 10.1007/s00423-012-0992-y. Epub 2012 Aug 24. PMID 22918605
- [Result] Yin Z, Fan X, Ye H, Yin D, Wang J. Short- and long-term outcomes after laparoscopic and open hepatectomy for hepatocellular carcinoma: a global systematic review and meta-analysis. Ann Surg Oncol. 2013 Apr;20(4):1203-15. doi: 10.1245/s10434-012-2705-8. Epub 2012 Oct 26. PMID 23099728